CLINICAL TRIAL: NCT04125797
Title: A Single Centre Comparison Study on Adhesion Properties of Three (3) Skin Adhesives on Healthy, Female, Adult Volunteers
Brief Title: Study on Adhesion Properties of Three Different Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambu A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CIS-015
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adhesive 1 (Active Comparator): This arm investigates one type of silicone adhesive (3M2475P) on adult female skin.
  Interventions: Other: Application of adhesive
- Adhesive 2 (Active Comparator): This arm investigates one type of silicone adhesive (RX1449P) on adult female skin.
  Interventions: Other: Application of adhesive
- Adhesive 3 (Active Comparator): This arm investigates one type of silicone adhesive (PS-1243) on adult female skin.
  Interventions: Other: Application of adhesive

INTERVENTIONS:
Other: Application of adhesive — Adhesive will be placed on the subjects skin below the bra. Placement of the adhesive will be randomized.

SUMMARY:
This clinical investigation is a single centre, double blinded, case control study in healthy adult females. This study will be conducted in private rooms at Gentofte Hospital (Hjerte-medicinsk Forskning, post 835, Kildegårdsvej 28, 2900 Hellerup).

The investigation centre will enroll 39 subjects including a 20% drop out within a four (4) months period. The subject will not be enrolled before approval of investigation protocol by the local ethics committee.

The subjects need to meet the inclusion and exclusion criteria to be included in this clinical investigation. Each volunteer enrolled in the investigation can only participate once in a procedure. The testing period for each subject will be minimum 72 hours.

The principal investigator's qualifications will be verified through his/her CV. The principal investigator is required to be a medical doctor with at least one year's experience in using similar medical adhesives (e.g. by being experienced in using electrodes where medical adhesives are included) and at least one year's experience with clinical research. In addition, the investigator must be trained in GCP before the study is initiated.

If any subject withdraws from the study, they will not be replaced as drop-out rate is included in the sample size.

Subjects must show up for two sessions, in the first session six adhesives will be placed below the subjects bra. The adhesives will be removed after minimum 72 hours at the second visit. While wearing the adhesives the subjects must keep the investigational area dry. 24, 48 and 72 hours after placement of the adhesives, the subject is asked to completed a questionnaire.

The eCRF must be completed for each subject that has signed the Informed consent form (ICF) and enrolled into this clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Female Healthy Volunteers.
* Age 18 - 40 years old.
* Willing to attend two scheduled visits
* Able to assess itch and adherence at 24h, 48h and 72h.
* Provide written informed consent.

Exclusion Criteria:

* Non-intact skin barrier (e.g. eczema, rash, cut, scar tissue, wound, etc.).
* History of inflammatory skin diseases (e.g. atopic dermatitis or psoriasis).
* History of contact allergy
* Swimming or engaging in sport activities causing sweat during study peri-od. v. Use of medication (e.g. corticosteroids) which could affect skin reactions.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Skin adhesion rating | Minimum 72 hours after application
  Rate of adhesion on a 5-point scale (no lift off the skin to deattached and completely off the skin)

SECONDARY OUTCOMES:
Itch | 24, 48 and 72 hours after adsive application
  Subject evaluation of itch during removal measured on visual analogue scale (0-10)
Ease of removal | Minimum 72 hours after application
  Ease of removal on 5-point scale (very difficult to very easy)
Pain during removal of adhesive | Minimum 72 hours after application
  Subject evaluation of pain during removal measured on visual analogue scale (0-10)
Rate of skin reaction | Minimum 72 hours after application
  Skin reaction rated on a scale from 0-7 (no evidence of irritation to strong reaction spreading beyond the application site)
Adhesive residue | Minimum 72 hours after application
  Adhesioe residue left on skin after removal of adhesive (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No